CLINICAL TRIAL: NCT07218250
Title: Piloting Single Session Consultation for Cancer (SSC-C) to Alleviate Distress Among Breast Cancer Patients
Brief Title: A Study of a One-Time Counseling Session to Help Reduce Depression, Anxiety, and Distress in People With Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: The City College of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-281
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: Counseling Session; Reduce Depression; Reduce Anxiety; Reduce Distress; 25-281
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSC-C - Single Session Consultation for Cancer (Experimental): will receive the study counseling
  Interventions: Behavioral: Single Counseling Session
- PPSB - Psychosocial Patient Support Booklet (Active Comparator): will receive an American Cancer Society booklet for review (and no counseling)
  Interventions: Other: American Cancer Society booklet

INTERVENTIONS:
Behavioral: Single Counseling Session — The one-time counseling session will be a problem-solving focused program that will try to strengthen the belief in the ability to manage the challenges of the cancer diagnosis and treatment
  Arms: SSC-C - Single Session Consultation for Cancer
Other: American Cancer Society booklet — called "After Diagnosis: A Guide for Patients and Families" for review. Again, this booklet includes information about cancer, living with cancer, making treatment decisions, talking to others about cancer, cancer treatment, and questions for the cancer care team. It will be given in person or by email.
  Arms: PPSB - Psychosocial Patient Support Booklet

SUMMARY:
The purpose of this study is to see if a Single Counseling Session for Cancer can help reduce psychosocial distress and improve quality of life in people with breast cancer who are waiting to receive ongoing counseling services (outpatient psychotherapy services). The Single Counseling Session for Cancer-which I will refer to as the "study counseling" during this call-is a one-session, 60-minute counseling program designed to reduce anxiety and depression symptoms in people with cancer who are waiting to receive outpatient psychotherapy services. The researchers will look at whether the study counseling is effective in participants and practical (feasible) for them to complete.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have pathologically confirmed breast cancer (per EMR).
* Patient with localized or advanced cancer (per EMR).
* Patient is on a waitlist of at least 2 weeks or more for MSK Counseling Center intake and will not complete a Counseling Center intake prior to intervention (these patients will be replaced) (per EMR, patient's care team, or self-report).
* Has no current active or passive suicidal ideation (per self-report of PHQ-9, Item 9: Thoughts that you would be better off dead, or of hurting yourself).
* Female (per EMR)
* Age ≥ 18 (per EMR)
* English fluency - Per self-report: How well do you speak English?
* Agrees to be audio-recorded (per self-report) NOTE: Participants who report Very well are considered fluent.
* Lives in New York, New Jersey, or Connecticut (per self-report).
* Has no significant psychiatric disturbance sufficient to preclude completion of the assessment measures, interview, or informed consent (i.e., acute psychiatric symptoms which require urgent or extended individual treatment) (per EMR, patient's care team, or study team).
* Has no presence of cognitive impairment disorder (i.e., delirium or dementia) sufficient to preclude meaningful informed consent and/or data collection (per EMR, patient's care team, or per self-report of BOMC cognitive test).
* Has no current active or passive suicidal ideation (per item 9 of the PHQ-9 and the CSSRS).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Enrollment: 20 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Acceptability (SSC-C participants) | up to 3 months
  Participants will complete a satisfaction survey after completing the SSC-C intervention. A 5-item, investigator- initiated, face-valid satisfaction survey will assess the degree with which participant found SSC-C helpful in developing an action plan to address their concerns, their perceived utility of the action plan, the degree with which they believe they will use the action plan, their motivation to do so, and the extent to which they will recommend SSC-C to other patients.
Acceptability (PPSB participants) | up to 3 months
  Participants will complete a satisfaction survey after receiving PPSB intervention materials. A 6-item, investigator- initiated, face-valid satisfaction survey will assess the degree with which participants found PPSB intervention helpful in developing an action plan to address their concerns, their perceived utility of the booklet, the degree with which they believe they will use the booklet, their motivation to do so, and the extent to which they will recommend the booklet materials to other patients.

SECONDARY OUTCOMES:
Psychosocial distress | up to 3 months
  The Hospital Anxiety and Depression Scale (HADS) will assess symptoms of anxiety (7 items, range 0-21) and depression (7 items, range 0-21).

CONTACTS AND LOCATIONS:
Overall Officials: Devika Jutagir, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm